CLINICAL TRIAL: NCT05360394
Title: A Prospective, Randomized Controlled Trial of Stent Graft and Drug Coated Balloon Treatment for Recurrent Cephalic Arch Stenosis in Dysfunctional Arteriovenous-venous Fistula
Acronym: PREDATOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2021/2044
Record Dates: First submitted 2022-04-26; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Neointimal Hyperplasia; Dialysis Access Malfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCB Only (Active Comparator): Cephalic arch stenosis is first treated with conventional plain balloon angioplasty. Once treated adequately (<30% residual stenosis), CAS will be treated with PCB angioplasty.
  Interventions: Device: Paclitaxel Coated Balloon
- Stent Graft and PCB angioplasty of stent edges (Experimental): CAS is first treated with conventional plain balloon angioplasty. Once treated adequately (<30% residual stenosis), CAS will be treated with PCB first to avoid geographical miss. After which, stent graft will be deployed. Length of PCB shall be long enough to cover stent edges.
  Interventions: Device: Paclitaxel Coated Balloon and Stent Graft

INTERVENTIONS:
Device: Paclitaxel Coated Balloon — CAS treated with PCB only
  Arms: PCB Only
Device: Paclitaxel Coated Balloon and Stent Graft — CAS treated with PCB first before deployment of stent graft
  Arms: Stent Graft and PCB angioplasty of stent edges

SUMMARY:
Arteriovenous Fistula (AVF) is a surgically created circuit used for hemodialysis in patient with End Stage Renal Disease (ESRD). A functioning dialysis vascular access is critical to the delivery of life-saving hemodialysis (HD) treatment for these patients. Unfortunately, neointimal hyperplasia frequently occurs within the dialysis vascular access, resulting in stenosis, poor flow and thrombosis with loss of function.

The cephalic vein forms the outflow conduit for radiocephalic (RC) and brachiocephalic (BC) AVF. At the perpendicular portion of the cephalic vein, the cephalic arch is often prone to developing hemodynamically significant stenosis. The prevalence of cephalic arch stenosis is reported to be 39% in brachiocepahlic and 2% in radiocephalic AVF.

The current gold standard therapy for treatment of AVF stenosis is plain balloon angioplasty (BA). Paclitaxel coated balloon (PCB) angioplasty has also been shown recently to be superior to plain BA in the treatment of stenosis in dialysis vascular access. By releasing paclitaxel, which is an anti-proliferation drug, locally into the vessel wall during balloon contact, it will blunt the acceleration of intimal hyperplasia response, resulting in improved primary patency after angioplasty.

The use of stent grafts for recurrent CAS has been demonstrated to increase patency of AVF compared to BA and bare stents. However, stent grafts are prone to edge restenosis that tend to occur within 5mm of each end of SG due to neointimal hyperplasia from the end of the stent migrating towards the center. We postulate that stent graft with PCB angioplasty of the stent edge is more effective than PCB alone in maintaining the patency of AVF with cephalic arch stenosis.

Therefore, we aim to perform a randomized controlled trial to compare the 6-month unassisted patency rate of treatment of recurrent CAS with stent graft and PCB angioplasty of both stent edge versus PCB alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 90 years
* Patients who requires balloon angioplasty for dysfunctional arteriovenous fistula, can be de novo lesions or recurrent CAS stenosis within six months of interventions. Suitability will be determined with a baseline ultrasound assessment.
* Matured AVF, defined as being in use for at least 1 month prior to angioplasty
* Successful angioplasty of the underlying stenosis, defined as less than 30% residual stenosis on Digital Subtraction Angiography (DSA).

Exclusion Criteria:

* Patient unable to provide informed consent
* Thrombosed or partially thrombosed AVF
* Immature AVF
* Insignificant CAS defined as <50% stenosis and no clinical indicator such as high V pressure.
* Presence of central vein stenosis with more than 30% residual stenosis post-angioplasty
* Patient who had underwent stent placement within the CAS previously
* Patients who are allergic to both aspirin or clopidogrel
* Patient who are currently enrolled in other drug eluting balloon trials
* Sepsis or active infection
* Recent intracranial bleed or gastrointestinal bleed within the past 12 months.
* Allergy to iodinated contrast media, heparin or paclitaxel
* Pregnancy

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Primary Patency of Target Lesion (Cepahlic Arch) | 6-months post-op
  Freedom from any re-intervention at target lesion that is clinically driven or indicated on surveillance scan
Primary Patency of Access Circuit | 6-months post-op
  Percentage of patients who do not need to undergo another re-intervention at the dialysis access circuit

SECONDARY OUTCOMES:
Primary Patency of Target Lesion | 3 and 12 months post-op
  Percentage of patients who do not need to undergo another re-intervention at the target lesion
Primary Patency of Access Circuit | 3 and 12 months post-op
  Freedom from any re-intervention that is clinically driven or indicated on surveillance scan
Assisted Primary Patency of Target Lesion | 3 and 12 months post-op
  Percentage of patients who do not need to undergo another thrombolysis or thrombectomy at target lesion.
Assisted Primary Patency of Access Circuit | 3 and 12 months post-op
  Percentage of patients who do not need to undergo another thrombolysis or thrombectomy at dialysis access circuit
Secondary Patency | 3 and 12 months post-op
  Percentage of patients who will not need creation of a new AVF or an alternative dialysis access site.
Time taken to next intervention | 12-months post-op
Number of repeat interventions to target lesion | 6 and 12 months post-op
Number of repeat interventions to maintain access circuit | 6 and 12 months post-op
Rate of late lumen loss of the cephalic arch, proximal and distal stent edge | 12 months post-op
Complication Rate | 1, 3, 6 and 12 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Tang Tjun Yip, Principal Investigator — Singapore General Hospital; Tan Ru Yu, Principal Investigator — Singapore General Hospital; Tay Kiang Hiong, Principal Investigator — Singapore General Hospital
Locations (2):
- Flinders Medical Center, Adelaide, Australia
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roy-Chaudhury P, Sukhatme VP, Cheung AK. Hemodialysis vascular access dysfunction: a cellular and molecular viewpoint. J Am Soc Nephrol. 2006 Apr;17(4):1112-27. doi: 10.1681/ASN.2005050615. PMID 16565259
- [Background] Rajan DK, Clark TW, Patel NK, Stavropoulos SW, Simons ME. Prevalence and treatment of cephalic arch stenosis in dysfunctional autogenous hemodialysis fistulas. J Vasc Interv Radiol. 2003 May;14(5):567-73. doi: 10.1097/01.rvi.0000071090.76348.bc. PMID 12761309
- [Background] Trerotola SO, Roy-Chaudhury P, Saad TF. Drug-Coated Balloon Angioplasty in Failing Arteriovenous Fistulas: More Data, Less Clarity. Am J Kidney Dis. 2021 Jul;78(1):13-15. doi: 10.1053/j.ajkd.2021.02.331. Epub 2021 May 8. No abstract available. PMID 33975757
- [Background] Irani FG, Teo TKB, Tay KH, Yin WH, Win HH, Gogna A, Patel A, Too CW, Chan SXJM, Lo RHG, Toh LHW, Chng SP, Choong HL, Tan BS. Hemodialysis Arteriovenous Fistula and Graft Stenoses: Randomized Trial Comparing Drug-eluting Balloon Angioplasty with Conventional Angioplasty. Radiology. 2018 Oct;289(1):238-247. doi: 10.1148/radiol.2018170806. Epub 2018 Jul 24. PMID 30040057
- [Background] Swinnen JJ, Hitos K, Kairaitis L, Gruenewald S, Larcos G, Farlow D, Huber D, Cassorla G, Leo C, Villalba LM, Allen R, Niknam F, Burgess D. Multicentre, randomised, blinded, control trial of drug-eluting balloon vs Sham in recurrent native dialysis fistula stenoses. J Vasc Access. 2019 May;20(3):260-269. doi: 10.1177/1129729818801556. Epub 2018 Sep 18. PMID 30227772
- [Background] Shemesh D, Goldin I, Zaghal I, Berlowitz D, Raveh D, Olsha O. Angioplasty with stent graft versus bare stent for recurrent cephalic arch stenosis in autogenous arteriovenous access for hemodialysis: a prospective randomized clinical trial. J Vasc Surg. 2008 Dec;48(6):1524-31, 1531.e1-2. doi: 10.1016/j.jvs.2008.07.071. Epub 2008 Oct 1. PMID 18829240
- [Background] Rajan DK, Falk A. A Randomized Prospective Study Comparing Outcomes of Angioplasty versus VIABAHN Stent-Graft Placement for Cephalic Arch Stenosis in Dysfunctional Hemodialysis Accesses. J Vasc Interv Radiol. 2015 Sep;26(9):1355-61. doi: 10.1016/j.jvir.2015.05.001. PMID 26074027
- [Background] Ginsburg M, Lorenz JM, Zivin SP, Zangan S, Martinez D. A practical review of the use of stents for the maintenance of hemodialysis access. Semin Intervent Radiol. 2015 Jun;32(2):217-24. doi: 10.1055/s-0035-1549844. No abstract available. PMID 26038628